CLINICAL TRIAL: NCT05628077
Title: Doctor of Medical Sciences
Brief Title: Prevalence and Risk Factors for Pain and Related Adverse Reactions Among Breast Cancer Survivors on Aromatase Inhibitors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Yi Feng, MD, Dr, Peking University People's Hospital
Other Study IDs: yifeng
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer; Aromatase Inhibitors; Endocrine Therapy; Pain; Anxiety; Depression; Sleep
MeSH Terms: conditions — Breast Neoplasms; Pain; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PAIN
  Interventions: Other: No intervention
- NO PAIN
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
We obtained the occurrence of pain sensation, pain mood, sleep, etc. during endocrine therapy in breast cancer patients through telephone follow-up, and analyzed risk factors through artificial intelligence

ELIGIBILITY:
Inclusion Criteria:

- Breast cancer survivors on aromatase inhibitors

Exclusion Criteria:

* Advanced breast cancer

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: I-III Breast cancer survivors on aromatase inhibitors
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-12-30 (Actual); Primary Completion 2023-03-20 (Estimated); Study Completion 2023-04-20 (Estimated)

PRIMARY OUTCOMES:
Prevalence and risk factors for pain and related adverse reactions among breast cancer survivors on aromatase inhibitors | 2022-10 ---2023-03

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People'S Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided